CLINICAL TRIAL: NCT00391170
Title: Pilot Study of Topical Dexamethasone 0.01% Solution for Prevention of Oral Chronic Graft Versus Host Disease
Brief Title: Dexamethasone to Prevent Oral Chronic Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 070005; 07-H-0005
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-02-24

CONDITIONS: Graft vs Host Disease
Keywords: Oral Chronic GVHD; Topical Dexamethasone; Tissue Markers; Salivary Proteomics; Quality of Life; Oral Chronic Graft Versus Host Disease; Oral Pain; Mouth Pain
MeSH Terms: conditions — Graft vs Host Disease | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone oral rinse in stem cell transplant participants (Experimental): Dexamethasone 0.01% (0.5mg/5 mL) oral rinse solution in post allogeneic hematopoietic stem cell transplant participants. Rinse oral cavity three times daily for two minutes with ten milliliters then expectorate. Complete for three months duration.
  Interventions: Drug: Topical Dexamethasone
- Placebo oral rinse in stem cell transplant participants (Placebo Comparator): Placebo oral rinse in post allogeneic hematopoietic stem cell transplant participants. Rinse oral cavity three times daily for two minutes with ten milliliters then expectorate. Complete for three months duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical Dexamethasone — dexamethasone 0.01%
  Arms: Dexamethasone oral rinse in stem cell transplant participants
Drug: Placebo — Placebo
  Arms: Placebo oral rinse in stem cell transplant participants

SUMMARY:
This study will determine if a dexamethasone mouth rinse can reduce the risk of developing oral chronic graft-versus-host disease (cGVHD) in patients who have undergone a bone marrow (stem cell) transplant procedure. cGVHD is a common complication of stem cell transplantation, resulting from the donor cells attacking the transplant recipient's tissues. In oral cGVHD, the tissues in the mouth are damaged, causing painful mouth sores. Dexamethasone is a corticosteroid that is commonly used to treat inflammation. It is the only corticosteroid available that can be used as a mouth rinse.

Patients 12 years of age or older who have received a stem cell transplant may be eligible to participate if they are enrolled within 70 to 90 days of their transplant. Candidates are screened with a medical history and oral exam.

Participants are randomly assigned to receive either the dexamethasone rinse or a placebo (a solution that looks and tastes like the dexamethasone rinse but has no active medication). They undergo the following procedures:

Treatment with the study solution. Patients rinse their mouth with the dexamethasone solution or placebo three times a day for 3 months.

Clinic visits before starting treatment and at 1, 2 and 3 months after starting the study drug for the following procedures:

* Oral exam (before starting treatment and at each visit).
* Photographs of the mouth (before starting treatment and at 3 months).
* Biopsy from inside the cheek (before starting treatment). The inside of the cheek is numbed and a small piece of tissue is removed for examination by a pathologist.
* Saliva sample collection (before starting treatment).
* Blood draw (before starting treatment and at each visit).
* Quality-of-life questionnaires (before starting treatment and at 3 months).
* Questionnaire to assess level of dry mouth and mouth pain (before starting treatment and at each visit).
* Review of medications (at each visit).
* ACTH stimulation test to evaluate adrenal gland function (at 3 months). Patients are given an injection of a drug called "ACTH" or "cosyntropin" which is a version of a hormone normally produced by the pituitary gland. Blood samples are drawn before the injection and at 30 and 60 minutes after the injection to measure levels of the hormone cortisol.

After treatment ends, participants are contacted by telephone every month for 6 months to report any symptoms of cGVHD, and they return to the clinic at 6 months for a final evaluation.

DETAILED DESCRIPTION:
Prevention of oral chronic graft versus host disease (GVHD) by topical agents is an attractive strategy because it would potentially avoid the adverse effects associated with systemic immunosuppression. Topically administered dexamethasone solution is a commonly used agent for the prophylaxis of oral inflammatory conditions including GVHD. However, the efficacy and systemic effects of topically administered dexamethasone solution are unknown. We therefore propose this trial designed to evaluate the efficacy and safety of topical dexamethasone solution for prevention of oral chronic GVHD in stem cell transplant recipients.

This pilot phase II study will follow a randomized, double-blind, placebo controlled, parallel group design. Consenting subjects who have undergone hematopoietic stem cell transplantation at the NIH Clinical Center and the surrounding transplant clinics will be randomized 50/50 to receive dexamethasone 0.01% solution or placebo as an oral rinse for 3 months starting 90-100 days post-transplant. Subjects will be evaluated monthly after the start of intervention. Diagnostic and research evaluations will include a complete oral examination, oral mucosal biopsy prior to the beginning of the intervention (day -7) and at the time of development of oral chronic GVHD or at the completion of intervention in the absence of clinical GVHD. We will measure serum dexamethasone levels and perform short cosyntropin (ACTH stimulation) test at the end of the 3 months of intervention or onset of clinically significant GVHD.

The primary objective of the study is to evaluate the safety and efficacy of topical dexamethasone 0.01% solution used as an oral rinse for prevention of oral chronic GVHD. Our primary endpoint will be the proportion of subjects that develop clinically significant (severity score 3 or higher) oral chronic GVHD after three months.

Secondary objectives will include the impact of oral chronic GVHD on the quality of life, characterization of the changes in tissue and salivary biomarkers associated with development of oral graft versus host disease, and measures of the effects of topical dexamethasone on hypothalamo-pituitary-adrenal axis. Secondary outcomes will include oral cavity specific quality of life as measured by Oral Health Impact Profile (OHIP)-14 questionnaire, oral discomfort levels, improvement in general quality of life scores, and severity of oral chronic GVHD as measured by the site-specific GVHD scoring system.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. History of allogeneic hematopoietic stem cell transplantation within 60-90 days of enrollment.
  2. Age 12 or older.
  3. Ability to rinse and expectorate study medication rather than swallow it.
  4. Ability and willingness to come to Clinical Center for follow-up appointments and at the time of development of symptoms/signs suggestive of oral GVHD.

EXCLUSION CRITERIA:

1. Clinically significant oral chronic GVHD at the time of the screening.
2. Active viral or fungal infection involving oral cavity not resolving by day 90.
3. Platelet count less than 20,000/ml at the time of the screening appointment.
4. Life expectancy less than 4 months at the time of enrollment.
5. Documented hypersensitivity to dexamethasone.
6. Pregnancy or lactation.
7. Inability to understand the investigational nature of the study.
8. Inability to provide informed consent.

Ages: 12 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-11-24 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Clara, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chakrabarti S, Childs R. Allogeneic immune replacement as cancer immunotherapy. Expert Opin Biol Ther. 2003 Oct;3(7):1051-60. doi: 10.1517/14712598.3.7.1051. PMID 14519070
- [Background] Tykodi SS, Warren EH, Thompson JA, Riddell SR, Childs RW, Otterud BE, Leppert MF, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation for metastatic renal cell carcinoma after nonmyeloablative conditioning: toxicity, clinical response, and immunological response to minor histocompatibility antigens. Clin Cancer Res. 2004 Dec 1;10(23):7799-811. doi: 10.1158/1078-0432.CCR-04-0072. PMID 15585611
- [Background] Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2003 Apr;9(4):215-33. doi: 10.1053/bbmt.2003.50026. PMID 12720215
- [Background] Thongprasom K, Luengvisut P, Wongwatanakij A, Boonjatturus C. Clinical evaluation in treatment of oral lichen planus with topical fluocinolone acetonide: a 2-year follow-up. J Oral Pathol Med. 2003 Jul;32(6):315-22. doi: 10.1034/j.1600-0714.2003.00130.x. PMID 12787037
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-H-0005.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 62 participants were consented. 54 participants started the study and 8 participants were screen failure.
Groups:
- Dexamathasone Oral Rinse in Stem Cell Transplant Participants: Dexamethasone 0.01% (0.5mg/5 mL) oral rinse solution in post allogeneic hematopoietic stem cell transplant participants. Rinse oral cavity three times daily for two minutes with ten milliliters then expectorate. Complete for three months duration.
Period: Overall Study
Arm/Group | Dexamathasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
Started | 27 | 27
Completed | 21 | 23
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamathasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 8 | 9 | 17
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Participants That Developed Severity Score 3 or Higher Oral Chronic Graft Versus Host Disease (GVHD).
Description: Participants that developed clinically significant (severity score 3 or higher) oral chronic graft versus host disease (GVHD) within 90 days of initiating treatment. Oral chronic GVHD is defined by Lichen Planus (Oral GVHD) Severity Scale (Thongprasom et al., 2003).
  Score 5: White striae with erosive area > 1 cm^2 Score 4: White striae with erosive area < 1 cm^2 Score 3: White striae with erythematous area > 1 cm^2 Score 2: White striae with erythematous area < 1 cm^2 Score 1: Mild white striae only Score 0: No lesions, normal mucosa
Time Frame: Day 90
Population: Stem cell transplant participants who started the dexamethasone oral rinse. An intention to treat analysis will be conducted as the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
Number analyzed (Participants) | 27 | 27
Participants | 7 | 4

2. Secondary Outcome: Participants With Chronic Oral Graft Versus Host Disease (GVHD) Based on Severity Scores
Description: Participants that developed oral chronic graft versus host disease (GVHD) within 90 days of initiating treatment. Oral chronic GVHD is defined by Lichen Planus (Oral GVHD) Severity Scale (Thongprasom et al., 2003).
  Score 5: White striae with erosive area > 1 cm^2 Score 4: White striae with erosive area < 1 cm^2 Score 3: White striae with erythematous area > 1 cm^2 Score 2: White striae with erythematous area < 1 cm^2 Score 1: Mild white striae only Score 0: No lesions, normal mucosa
Time Frame: Day 90
Population: Stem cell transplant participants who started and completed the study intervention. Three participant were nonevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
Number analyzed (Participants) | 25 | 26
Participants
  Score of 0 | 17 | 19
  Score = 1 | 1 | 1
  Score = 2 | 0 | 2
  Score = 3 and > | 7 | 4

3. Secondary Outcome: Participants With Systemic Absorption of Topical Dexamethasone
Description: Participants with systemic absorption of topical dexamethasone based on plasma dexamethasone level < 30 ng/dL.
Time Frame: 3 months
Population: Stem cell transplant participants who started the dexamethasone oral rinse and completed dexamethasone blood draw at 3 month follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
Number analyzed (Participants) | 22 | 23
Participants | 1 | 0

4. Secondary Outcome: Participants With Suppressed Adrenal Cortical Function Due to Topical Dexamethasone
Description: Number of participants who are not on systemic steroids with suppressed adrenal cortical function after completing study intervention phase (3 month) based on serum morning cortisol levels.
Time Frame: 3 months
Population: Stem cell transplant participants who started the dexamethasone oral rinse and completed serum cortisol levels at 3 months follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
Number analyzed (Participants) | 20 | 19
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were assessed during clinic visits
Arm/Group | Dexamethasone Oral Rinse in Stem Cell Transplant Participants | Placebo Oral Rinse in Stem Cell Transplant Participants
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/27
Other Adverse Events (participants affected / at risk) | 13/27 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Oral Rinse in Stem Cell Transplant Participants (N=27) | Placebo Oral Rinse in Stem Cell Transplant Participants (N=27)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Oral Rinse in Stem Cell Transplant Participants (N=27) | Placebo Oral Rinse in Stem Cell Transplant Participants (N=27)
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Dry mouth (Gastrointestinal disorders) | 4 | 11
Oral pain (Gastrointestinal disorders) | 3 | 8
fatigue (General disorders) | 1 | 5
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Dizziness (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT00391170/Prot_SAP_000.pdf